CLINICAL TRIAL: NCT00229619
Title: A Pilot Study of Recombinant Humanized Anti- Cluster of Differentiation Antigen 20 (Anti-CD20) Antibody (Rituximab) in Patients With Moderate Aplastic Anemia, Pure Red Cell Aplasia, or Diamond Blackfan Anemia
Brief Title: Rituximab to Treat Moderate Aplastic Anemia, Pure Red Cell Aplasia, or Diamond Blackfan Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Adrian Wiestner, M.D., NHLBI Senior Investigator, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050244; 05-H-0244 (Other: NIH NHLBI)
Record Dates: First submitted 2005-09-29; First posted 2005-09-29 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Anemia, Aplastic; Red-Cell Aplasia, Pure; Anemia, Diamond-Blackfan
Keywords: rituxan; Immunosuppression; Bone Marrow Failure; Monoclonal Antibody Therapy; Diamond Blackfan Anemia (DBA); T -Cells; B-Cells; Hematopoiesis; Moderate Aplastic Anemia (MAA); Diamond-Blackfan Anemia; DBA; Pure Red Cell Aplasia; PRCA
MeSH Terms: conditions — Anemia, Aplastic; Red-Cell Aplasia, Pure; Anemia, Diamond-Blackfan; Bone Marrow Failure Disorders | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Rituxan) (Experimental): This is a non-randomized, off label, pilot study of humanized anti CD20 rituximab (Rituxan®) in patients with moderate aplastic anemia, pure red cell aplasia or Diamond-Blackfan anemia who have either failed to respond to at least one prior course of immunosuppressive therapy (PRCA/DBA patients only)or who have relapsed disease after prior immunosuppressive therapy (PRCA/DBA patients only).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab (Rituxan) 375mg/m2 intravenous infusion. The infusion will be once every week for a total of 4 doses.
  Other Names: Rituxan

SUMMARY:
This study will test whether the immune-suppressing drug rituximab can increase blood counts and reduce the need for transfusions in patients with moderate aplastic anemia, pure red cell aplasia, or Diamond Blackfan anemia. These are rare and serious blood disorders in which the immune system turns against bone marrow cells, causing the bone marrow to stop producing red blood cells in patients with pure red cell aplasia and Diamond Blackfan anemia, and red blood cells, white blood cells and platelets in patients with aplastic anemia. Rituximab is a laboratory-made monoclonal antibody that recognizes and destroys white blood cells called lymphocytes that are responsible for destroying bone marrow cells in these diseases. The drug is currently approved by the Food and Drug Administration for treating patients with B-cell non-Hodgkin lymphoma, a disease of white blood cells.

DETAILED DESCRIPTION:
This study will test whether the immune-suppressing drug rituximab can increase blood counts and reduce the need for transfusions in patients with moderate aplastic anemia, pure red cell aplasia, or Diamond Blackfan anemia. These are rare and serious blood disorders in which the immune system turns against bone marrow cells, causing the bone marrow to stop producing red blood cells in patients with pure red cell aplasia and Diamond Blackfan anemia, and red blood cells, white blood cells and platelets in patients with aplastic anemia. Rituximab is a laboratory-made monoclonal antibody that recognizes and destroys white blood cells called lymphocytes that are responsible for destroying bone marrow cells in these diseases. The drug is currently approved by the Food and Drug Administration for treating patients with B-cell non-Hodgkin lymphoma, a disease of white blood cells.

Participants receive four doses of rituximab, once a week for 4 weeks through a needle in an arm vein. The infusion rate depends on how well the patient tolerates the drug. The first infusion usually takes 4 to 6 hours and the rest take 3 to 4 hours. The first and fourth infusions are given at NIH; the second and third may be given at NIH or by a patient's referring doctor. Patients who respond to rituximab but then relapse may receive one additional course of four doses. Patients may continue with transfusions and their current medications, including growth factors (e.g., Epogen and Neupogen) while on study, but may have to stop taking immunosuppressive drugs, such as prednisone or cyclosporine. Patients who must start another immunosuppressive medication are taken off rituximab and followed for safety with clinic visits one week and then once a month for 6 months after the first dose of rituximab.

Patients have a blood test once a week while receiving rituximab to evaluate blood counts. After treatment is completed, patients are evaluated once a month until 6 months, then once a year until 3 years to monitor the response to treatment and any drug side effects. Patients are evaluated at NIH for the 3- and 6-month visits and the annual visits. They may be seen at NIH or by their referring doctors for the 1-, 2-, 4- and 5-month visits. A blood test is done at every visit, and a bone marrow aspiration and biopsy are done at the 3-month visit (and when clinically needed to evaluate the effect of rituximab on bone marrow cells).

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of acquired moderate aplastic anemia defined as aplastic anemia (hypocellular bone marrow) and no evidence for an underlying disease process and depression of at least two out of three blood counts below these values:

* Absolute neutrophil count (ANC) equal to or less than l200/mm(3)
* platelet count equal to or less than 70,000/mm(3)
* anemia with hemoglobin equal to or less than 8.5 g/dl or absolute reticulocyte count equal to or less than 60,000/mm(3) in transfusion-dependent patients but not fulfilling the criteria for severe disease defined by bone marrow cellularity less than 30% (excluding lymphocytes) and depression of at least two of the three peripheral counts:
* ANC equal to or less than 500/ul
* platelet count equal to or less than 20,000/ul
* reticulocyte count less than 60,000/ul

Or

Diagnosis of pure red cell aplasia or Diamond Blackfan anemia requiring red blood cell (RBC) transfusions

Pure red cell aplasia is defined by

* anemia,
* reticulocytopenia (reticulocyte count equal to or less than 50,000/ mm(3))
* and absent or decreased marrow erythroid precursors

Diamond Blackfan anemia is defined by

* anemia,
* reticulocytopenia (reticulocyte count equal to or less than 50,000/ mm(3))
* and absent or decreased marrow erythroid precursors diagnosed at an early age

Because this population is prone to dry bone marrow aspirates, subjects from whom sufficient bone marrow cannot be collected for the evaluation of cellularity will not be excluded provided they meet all other inclusion criteria based on peripheral blood counts.

Pure Red cell Aplasia and Diamond Blackfan patients must be age greater than or equal to 2 years old and weight greater than 12 kg; Moderate Aplastic anemia patients must be age greater than or equal to 18.

Refractory to at least 1 course of immunosuppressive therapy or relapsed disease after prior immunosuppressive therapy (PRCA/DBA patients only).

Patients or their parent(s)/responsible guardian(s) must be able to comprehend and be willing to sign an informed consent.

EXCLUSION CRITERIA:

Current diagnosis of Fanconi's anemia or other congenital bone marrow failure syndromes except for DBA

History of a cytogenetic abnormality indicating myelodysplasia (MDS)

Active infection not adequately responding to appropriate therapy

HIV positivity

Positive anti- hepatitis B core antibody (antiHBc) or HBsAG

History of clinically significant arrhythmia

Known anaphylaxis or immunoglobulin E (IgE) mediated hypersensitivity to murine proteins or to any component of this product.

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within the next month is likely

Potential subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible.

History of recent or ongoing B19 parvovirus infection

Psychiatric, affective, or other disorder that may compromise the ability to give informed consent or to cooperate in a research study.

Pregnancy or lactation or unwillingness to take contraceptives

Participation in any other investigational drug trial or exposure to other investigational agents (other than hematopoietic growth factors) within 30 days of study entry. Use of low dose immunosuppressive agents may continue at the PIs discretion provided that the patient has been taking this drug for at least 3 months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Martyr, MD, Principal Investigator — NIH National Heart, Lung, and Blood Institute
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wang J, Wiley JM, Luddy R, Greenberg J, Feuerstein MA, Bussel JB. Chronic immune thrombocytopenic purpura in children: assessment of rituximab treatment. J Pediatr. 2005 Feb;146(2):217-21. doi: 10.1016/j.jpeds.2004.09.004. PMID 15689912
- [Background] Gottenberg JE, Guillevin L, Lambotte O, Combe B, Allanore Y, Cantagrel A, Larroche C, Soubrier M, Bouillet L, Dougados M, Fain O, Farge D, Kyndt X, Lortholary O, Masson C, Moura B, Remy P, Thomas T, Wendling D, Anaya JM, Sibilia J, Mariette X; Club Rheumatismes et Inflammation (CRI). Tolerance and short term efficacy of rituximab in 43 patients with systemic autoimmune diseases. Ann Rheum Dis. 2005 Jun;64(6):913-20. doi: 10.1136/ard.2004.029694. Epub 2004 Nov 18. PMID 15550531
- [Background] Edwards JC, Szczepanski L, Szechinski J, Filipowicz-Sosnowska A, Emery P, Close DR, Stevens RM, Shaw T. Efficacy of B-cell-targeted therapy with rituximab in patients with rheumatoid arthritis. N Engl J Med. 2004 Jun 17;350(25):2572-81. doi: 10.1056/NEJMoa032534. PMID 15201414
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-H-0244.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Treated Subjects: Rituximab will be given to moderate aplastic anemia (MAA), pure red cell aplasia or Diamond Blackfan anemia subjects. Rituxmiab will be given to evaluate if these bone marrow failure syndrome subjects will have an immune response to the intervention. The subjects will receive 375 mg/ meters squared of rituximab which will be infused intravenously once evey week for a total of 4 doses.
Period: Overall Study
Arm/Group | Rituximab Treated Subjects
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Rituximab Subjects: Rituximab will be given to moderate aplastic anemia (MAA), pure red cell aplasia or Diamond Blackfan anemia subjects. Rituxmiab will be given to evaluate if these bone marrow failure syndrome subjects will have an immune response to the intervention. The subjects will receive 375 mg/ meters squared of rituximab which will be infused intravenously once evey week for a total of 4 doses.
Arm/Group | Rituximab Subjects
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Response to Rituximab
Description: Rituximab will be given to moderate aplastic anemia (MAA), pure red cell aplasia or Diamond Blackfan anemia subjects. Rituxmiab will be given to evaluate if these bone marrow failure syndrome subjects will have an immune response to the intervention. The subjects will receive 375 mg/ meters squared of rituximab which will be infused intravenously once evey week for a total of 4 doses.
  Primary endpoint will determine immune response by evaluating changes in peripheral blood counts (platelets, absolute neutrophil count, reticulocyte count, hemoglobin) and transfusion requirements at 6 months. The response wil be will be categorized as complete, partial or no response. Subjects will be categorized as complete responders if their blood counts return to normal. Subjects will categorized as partial responders if there is an improvement in 2 or 3 of the depressed baseline blood counts.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Rituximab Subjects
Number analyzed (Participants) | 11
participants
  Complete response | 0
  Partial response | 2
  No Response | 9

2. Secondary Outcome: Response Assessment at 3 Months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab (Rituxan)
Number analyzed (Participants) | 11
Participants
  Complete response | 0
  Partial response | 1
  No response | 10

3. Secondary Outcome: Response Rates at 12 Months (After the First Dose of Study Med)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Treated Subjects
Number analyzed (Participants) | 11
Participants
  Complete response | 0
  Partial response | 3
  Relapse after response | 1
  No response | 7

ADVERSE EVENTS:
Arm/Group | Rituximab Subjects
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Subjects (N=11)
Acidosis (Metabolism and nutrition disorders) | 1
Infection with normal ANC (Infections and infestations) | 1
right popliteal artery occlusion (Vascular disorders) | 1
Abdominal abscess (Infections and infestations) | 1
anemia (Blood and lymphatic system disorders) | 1 — symptomatic anemia
skin breakdown (Skin and subcutaneous tissue disorders) | 1 — Wound complication, non-infectious
Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Subjects (N=11)
Bleeding (Blood and lymphatic system disorders) | 1
Bruising (Blood and lymphatic system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cytokine release syndrome/ acute infusion reaction (General disorders) | 1
Pain (General disorders) | 2 — Localized pain, line insertion site
Serum sickness (Immune system disorders) | 1
Fatigue (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Mouth sores (Gastrointestinal disorders) | 1
Headache (General disorders) | 1
arrythmia (Cardiac disorders) | 1 — EKG changes
Mild swelling of extremity (Cardiac disorders) | 2
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 3
Pallor (General disorders) | 1
strep throat (Infections and infestations) | 1
dry, flaking skin temporal area (Skin and subcutaneous tissue disorders) | 2
Lymph node (Immune system disorders) | 1 — anterior lymph node-supraclavicular
urinary frequency/ dysuria (Hepatobiliary disorders) | 1
infection (Strep viridans) (Infections and infestations) | 1
fever (General disorders) | 1
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 1
Decreased hemoglobin (Blood and lymphatic system disorders) | 1
Decreased lymphocytes (Blood and lymphatic system disorders) | 1
Decreased platelets (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Right foot ulcer (Skin and subcutaneous tissue disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Splenomegaly (Gastrointestinal disorders) | 1
Increased LFTs (Hepatobiliary disorders) | 1
Upper respiratory tract (Infections and infestations) | 1
Arthralgia (General disorders) | 1
tooth pain (General disorders) | 1
Lip. Pimple (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to slow accrual. Conclusions on efficacy limited by small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes